CLINICAL TRIAL: NCT03791346
Title: Outcome After Pancreatectomy for Neuroendocrine Tumor and Evaluation of the WHO 2017 Grading System: a Retrospective Multicentric Analysis of 138 Consecutive Patients.
Brief Title: Pancreatectomy for NET: External Evaluation of WHO 2017 Grading System
Acronym: PanTEN
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Department of digestive surgery, Carémeau Hospital, 30900, Nîmes, France (Unknown); Department of oncology, Carémeau Hospital, 30900, Nîmes, France (Unknown); Oncology - Institut du Cancer de Montpellier (ICM), Montpellier, France (Unknown); Digestive & Oncologic Surgery - Institut du Cancer de Montpellier (ICM), Montpellier, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0492
Record Dates: First submitted 2018-12-31; First posted 2019-01-02 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-12

CONDITIONS: Pancreatic Surgery
Keywords: neuroendocrine tumor; Survival; WHO 2017 grading system; pancreatectomy; Laparoscopy; Postoperative outcomes
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Aim: The aim of this study was to investigate the clinicopathological factors and to evaluate the prognostic accuracy of the new World Health Organization (WHO) 2017 grading system in pancreatic neuroendocrine tumor (PanNET) patients.

Methods: Data collected between 1997 and December 2017 were analyzed. Histological grading and staging was based on the WHO 2017 grading system. Outcome after surgery and predictors of overall survival (OS) and disease free survival (DFS) were evaluated.

ELIGIBILITY:
Inclusion criteria:

- patients with histologically proven neuroendocrine tumor located in pancreas who underwent pancreatic resection (by open, laparoscopic or robotic approach) even in case of distant metastasis at time of surgery, with no previous or concurrent malignancy.

Exclusion criteria:

- Patients with tumors diagnosed as adenocarcinoma with scattered neuroendocrine cells or with focal neuroendocrine component were excluded of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective review of collected data including all consecutive patients requiring a pancreatic resection for PanNET at 3 tertiary referral centers for pancreatic surgery in France, between December 1997 and December 2017. The 3 centers were Digestive Surgery Units of Montpellier, Nimes and Institute of Cancer at the University of Montpellier-Nimes.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 1997-01-01 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival at 5 years | 5 years
  Disease-free survival (percentage of patients without recurrence) at 5 years. Disease-free survival (DFS) (time from diagnosis to time of first radiological evidence of local, regional, or distant relapse, or death due to any cause)

SECONDARY OUTCOMES:
Overall survival at 5 years | 5 years
  Overall survival (OS) (time from diagnosis until death, regardless of cause)

CONTACTS AND LOCATIONS:
Overall Officials: REGIS SOUCHE, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France